CLINICAL TRIAL: NCT05822050
Title: An Open, Single Center, Non-randomized, Single Arm Clinical Study of Evaluating the Efficacy of Selinexor in the Maintenance Treatment of Peripheral T-cell Lymphomas (PTCL)
Brief Title: An Open, Single Center, Non-randomized, Single Arm Clinical Study of Evaluating the Efficacy of Selinexor in the Maintenance Treatment of PTCL
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Ou Bai, MD/PHD, The First Hospital of Jilin University, The First Hospital of Jilin University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PTCL-001
Record Dates: First submitted 2023-03-30; First posted 2023-04-20 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: PTCL Patients Who Achieved Complete Response From Frontline Treatment
MeSH Terms: interventions — selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low risk group (Experimental): 10 patients. Selinexor 60mg QW Oral 21days/cycle
  Interventions: Drug: Selinexor
- Medium/High risk group (Experimental): 10 patients. Selinexor 60mg QW Oral with Chemotherapy 21days/cycle
  Interventions: Drug: Selinexor

INTERVENTIONS:
Drug: Selinexor — XPO1 inhibitor

SUMMARY:
To evaluate the efficacy and safety of Selinexor maintenance therapy in PTCL patients who achieved complete response from frontline treatment, and to analyze the relationship between gene mutation in PTCL and disease prognosis and clinical features by using Next-generation sequencing (NGS) detection.

ELIGIBILITY:
Inclusion Criteria:

* Patients fully understand the study, voluntarily participate and sign the informed consent (ICF);
* Age range from 18 to 85 years old (including upper and lower limits);
* ECOG (Eastern Cooperative Oncology Group) score 0 ~ 2;
* PTCL confirmed by histopathology falls into one of the following subtypes according to the WHO classification standard revised in 2016:1) Peripheral T-cell lymphoma non-specific type (PTCL-NOS) 2) vascular immunoblastic T-cell lymphoma (AITL) 3) ALK+ systemic anaplastic large T-cell lymphoma (ALK+ALCL) 4) Alk-systemic anaplastic large T-cell lymphoma (ALK-AlCl) 5) extranasal NK/ T-cell lymphoma (NK/TCL)6) Other subtypes of PTCL that the researchers considered suitable for inclusion.
* Subjects achieved complete remission by radiographic assessment at mid-stage.
* Subjects must provide a written pathological/histological diagnosis report during the screening period and must agree to provide tumor tissue sections or tumor/lymph node tissue samples for central laboratory testing.
* Expected survival is at least 12 weeks.
* Patients must meet the following requirements for laboratory tests at screening time and have not received cell growth factor, platelet, or granulocyte infusion within 7 days prior to screening hematological evaluation.1) Neutrophil absolute value ≥1.5×109/L in subjects without bone marrow involvement and ≥1.0×109/L in subjects with bone marrow involvement;2) Hemoglobin ≥90g/L in subjects without bone marrow involvement (in the absence of red blood cell infusion within 14 days), hemoglobin ≥75g/L in subjects with bone marrow involvement;3) Platelets ≥75×109/L in subjects without bone marrow involvement and ≥50×109/L in subjects with bone marrow involvement;4) Serum total bilirubin ≤1.5× upper limit of normal (ULN) (total bilirubin ≤3×ULN if elevated bilirubin level is caused by lymphoma invading the liver);5) Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤2.5×ULN;If elevated AST and ALT are caused by lymphoma invading liver, both AST and ALT should be ≤5×ULN).6) Creatinine <1.5×ULN.
* Eligible patients (male and female) who are fertile must agree to use a reliable contraceptive method (hormonal or barrier method or abstinence) with their partner during the trial period and for at least 7 months after the last medication;Female patients of reproductive age must have had a negative blood pregnancy test within 14 days prior to inclusion.

Exclusion Criteria:

* Patients with leukemic PTCL (such as adult T-cell leukemia/lymphoma, etc.), or lymphoma leukemia stage (bone marrow examination lymphoma cell proportion ≥20%), or central nervous system (CNS) involvement, or complicated hemophagocytic syndrome.
* Allergic history to similar drugs and excipients of the study drug.
* Participated in other clinical studies and used the study drug within 4 weeks prior to the first administration of the study drug.
* The toxic reactions of previous antitumor therapy have not recovered, and there are still more than grade 1 toxic reactions, except hair loss and pigmentation.
* Impaired heart function or significant heart disease, including but not limited to: 1) myocardial infarction, congestive heart failure, viral myocarditis in the 6 months prior to screening;Heart disease with symptoms that require therapeutic intervention, such as unstable angina, arrhythmia, etc.;2) Cardiac function grade Ⅱ to Ⅳ (New York College of Cardiology Cardiac Function Grade NYHA);3) Echocardiographic examination of cardiac ejection fraction (EF) below 50% or below the lower limit of laboratory test value;
* Active hepatitis B (surface antigen positive with HBV-DNA titers higher than 2000IU/ml) or hepatitis C (HCV antibody positive with HCV ribonucleic acid (HCV RNA) titers higher than the upper limit of the study center's normal).
* History of severe autoimmune diseases and immunodeficiency, including positive human immunodeficiency virus (HIV) antibodies;Or other acquired or congenital immunodeficiency diseases;Or have a history of organ transplantation.
* History of other malignant tumors within 5 years (except cured basal cell carcinoma of the skin and carcinoma in situ of the cervix).
* Major surgery was performed within 6 weeks prior to screening or was expected to be performed during the study period.
* There are significant gastrointestinal disorders at the time of screening that may affect drug intake, transport or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, etc.).
* Uncontrolled hypertension (refers to patients with type 2 diabetes whose blood pressure still reaches the level 3 hypertension standard after antihypertensive treatment, with systolic blood pressure ≥180mmHg and/or diastolic blood pressure ≥110mmHg) or who cannot be controlled by oral hypoglycemic drugs and insulin therapy.
* History of active bleeding within 3 months prior to screening.
* History of mental illness or psychotropic substance abuse or dependence.
* Pregnant or lactating women.
* Other conditions considered inappropriate for participation in the study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival rate of 1 year (1y PFS rate) | 1 year from the start of selinexor treatment
  progression-free survival rate, defined as the proportion of patients who have not experience PFS events after one year from the date of start of selinexor treatment. PFS events is defined as the first documentation of relapse or progressive disease, death due to any cause, or receipt of subsequent systemic chemotherapy to treat residual or progressive peripheral T-cell lymphoma as determined by the investigator, whichever came first.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | from the date of start of selinexor to the end of study
  progression-free survival, defined as the time from the date of start of selinexor treatment to the date of first documentation of relapse or progressive disease, death due to any cause, or receipt of subsequent systemic chemotherapy to treat residual or progressive peripheral T-cell lymphoma as determined by the investigator, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Bethune Hospital of Jilin University, Changchun, Jilin, China